CLINICAL TRIAL: NCT05547373
Title: Developing and Piloting an Infection Prevention and Control Intervention to Reduce Hospital-acquired Infections in Cambodia and Lao PDR
Brief Title: Infection Prevention and Control Intervention to Reduce Hospital-acquired Infections
Acronym: IPC-HAI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University of Singapore (Other)
Collaborators: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Siyan Yi, Assistant Professor, National University of Singapore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RCP100737ITDC
Record Dates: First submitted 2022-09-13; First posted 2022-09-21 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Hospital-acquired Infections
Keywords: Infection control; Prevention; Hand hygiene; Healthcare workers; Low- and middle-income countries; Asia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): The investigators will select HCWs from the selected departments at the national hospitals, provincial hospitals, and district referral hospitals to participate in the pilot intervention. The participants will also include representatives from the Communicable Disease Control Department and the Department of Hospital Services of the Ministry of Health, the provincial hospitals, and the district referral hospitals in Cambodia and Lao PDR.
  Interventions: Behavioral: Infection prevention and control (IPC)

INTERVENTIONS:
Behavioral: Infection prevention and control (IPC) — The intervention will be developed by matching behavioral change components identified in the gap analysis stage with the intervention components extracted from a systematic review. The investigators will use the Behavior Change Wheel (BCW) model as a guide to design this infection control prevention and control intervention. In brief, the intervention development processes will follow eight steps based on the BCW. The steps will include defining the problem in behavioral terms, selecting the target behaviors, specifying the target behaviors, identifying what needs to change, identifying intervention functions, identifying policy categories, identifying behavior change techniques, and identifying the mode of delivery.

SUMMARY:
Hospital-acquired infections (HAIs) are significant public health issues, especially in low- and middle-income countries (LMICs). Hand hygiene and low-level disinfection of equipment (LLDE) practices among healthcare workers (HCWs) are essential to reduce HAIs. Various effective infection prevention and control (IPC) interventions to reduce HAI incidence have been developed. However, which interventions work effectively in LMICs has not been identified. The investigators aim to develop, pilot, and assess the feasibility and acceptability of an IPC intervention in Cambodia and the Lao People's Democratic Republic (PDR).

DETAILED DESCRIPTION:
This study consists of four phases guided by the Medical Research Council (MRC) framework. Three hospitals from each country will be selected. In Phase 1, the investigators will conduct a gap analysis of IPC implementation and practices among HCWs at each hospital through desk review, direct observation of hand hygiene and LLDE practices, in-depth interviews with HCWs, and key informant interviews with stakeholders. In Phase 2, the investigators will develop an IPC intervention based on results from Phase 1 and interventions selected from the literature review of IPC interventions in LMICs. In Phase 3, the investigators will pilot the developed intervention in the same hospitals selected in Phase 1. Finally, in Phase 4, the investigators will assess the feasibility and acceptability of the developed intervention among HCWs and stakeholders at the selected hospitals. The investigators will employ the MRC framework to develop and evaluate an intervention to reduce HAIs in both countries. The investigators will also use a theoretical framework to explore factors that are barriers and enablers for HCWs to improve hand hygiene compliance. With these approaches, the investigators will be able to develop a comprehensive intervention. Findings from this study would shed light on promising IPC interventions to reduce HAI incidence in Cambodia and Lao PDR. More importantly, the findings may be applied to other LMIC settings.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare workers working in the selected wards and of chosen hospitals
* Aged 18 years or above
* Working in the selected wards of the chosen hospitals for at least six months
* Being able and agreeing to provide informed consent to participate in the study

Exclusion Criteria:

- Interns and visiting healthcare workers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in hand hygiene compliance among health workers from baseline to endline | At endline (6 months after the intervention started)
  The investigators will calculate hand hygiene compliance by having the hand hygiene action of alcohol hand rub or hand washing using soap and water divided by the hand hygiene opportunity and multiple with 100.

SECONDARY OUTCOMES:
Perceived feasibility and acceptability of the infection prevention and control intervention among HCWs and stakeholders | At endline (6 months after the intervention started)
  The investigators will conduct a post-intervention qualitative evaluation to assess the feasibility and acceptability and identify challenges in implementing the infection prevention and control intervention following the Medical Research Council's framework.

CONTACTS AND LOCATIONS:
Locations (1):
- Khmer-Soviet Friendship Hospital, Phnom Penh, Cambodia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oy S, Saing CH, Ung M, Zahari M, Nouhak I, Kim S, Nagashima-Hayashi M, Khuon D, Koy V, Mam S, Sayasone S, Saphonn V, Yi S. Developing an infection prevention and control intervention to reduce hospital-acquired infections in Cambodia and Lao People's Democratic Republic: the HAI-PC study protocol. Front Public Health. 2023 Sep 20;11:1239228. doi: 10.3389/fpubh.2023.1239228. eCollection 2023. PMID 37799162